CLINICAL TRIAL: NCT00619866
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NBI-56418 in Subjects With Endometriosis
Brief Title: An Efficacy and Safety Study of Elagolix (NBI-56418) in Women With Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-56418-0702
Record Dates: First submitted 2008-01-24; First posted 2008-02-21 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-03

CONDITIONS: Endometriosis, Pain
Keywords: bone mineral density; Pelvic Pain; estradiol; NBI-56418
MeSH Terms: conditions — Endometriosis; Pain; Pelvic Pain | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo tablets once a day for 12 weeks. At the end of 12 weeks participants were re-randomized to receive one of the two doses of elagolix (150 mg or 250 mg) QD for 12 weeks.
  Interventions: Drug: placebo
- Elagolix 150 mg (Experimental): Participants received elagolix 150 mg tablets once a day for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 150 mg QD for an additional 12 weeks.
  Interventions: Drug: Elagolix
- Elagolix 250 mg (Experimental): Participants received elagolix 250 mg tablets once a day for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 250 mg for an additional 12 weeks.
  Interventions: Drug: Elagolix

INTERVENTIONS:
Drug: Elagolix — Elagolix tablets administered orally
  Other Names: NBI-56418; Orilissa™
  Arms: Elagolix 150 mg; Elagolix 250 mg
Drug: placebo — Placebo tablet administered orally
  Arms: Placebo

SUMMARY:
This study is designed to see how elagolix works compared to placebo in women with endometriosis and to see the effect, if any, on bone mineral density.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled parallel-group study to assess the efficacy and safety of elagolix at two dose levels administered once daily for up to 6 months. Participants will be randomized (1:1:1) to one of the following treatment groups for the first 12 weeks of dosing: 150 mg elagolix once daily (QD); 250 mg elagolix QD or placebo QD. Following 12 weeks of dosing, participants will continue in the study for an additional 12 weeks; participants randomized to elagolix will continue to receive their assigned dose and participants randomized to placebo will be re-randomized to receive one of the two doses of elagolix for 12 weeks in a double-blind fashion. Six weeks after the last dose of study drug at the end of Week 24, a follow-up visit will be performed (end of Week 30).

ELIGIBILITY:
Inclusion Criteria:

* Be female, aged 18 to 49 years, inclusive
* Have moderate to severe pelvic pain due to endometriosis
* Have been surgically (laparoscopy) diagnosed with endometriosis within the last 8 years and have recurrent or persistent endometriosis symptoms
* Have regular menstrual cycle
* Have a body mass index (BMI) of 18 to 36 kg/m², inclusive
* Agree to use two forms of non-hormonal contraception during the study

Exclusion Criteria:

* Are currently receiving gonadotropin-releasing hormone (GnRH) agonist or GnRH antagonist or have received any of these agents within 6 months of the start of screening
* Are currently receiving subcutaneous medroxyprogesterone acetate (DMPA-SC) or intramuscular medroxyprogesterone acetate (DMPA-IM) or have received any of these agents within 3 months of the start of screening
* Are currently using hormonal contraception or other forms of hormonal therapy or received such treatment within the last month
* Have had surgery for endometriosis within the last month
* Have had a hysterectomy or bilateral oophorectomy
* Are using systemic steroids on a chronic or regular basis within 3 months
* Have uterine fibroids ≥ 3 cm in diameter
* Have pelvic pain that is not caused by endometriosis
* Have unstable medical condition or chronic disease
* Have been pregnant within the last six months
* Currently breast feeding

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2008-02-19 (Actual); Primary Completion 2009-04-20 (Actual); Study Completion 2009-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 50 centers in the United States from February 2008 to August 2009.
Pre-assignment Details: Patients were randomized equally to oral elagolix 150 mg or 250 mg once daily, or placebo for 12 weeks. Thereafter, patients originally randomized to placebo were re-randomized to one of the two elagolix doses and patients originally randomized to elagolix continued their assigned dose for an additional 12 weeks.
Groups:
- Placebo: Participants received placebo tablets once a day (QD) for 12 weeks. At the end of 12 weeks participants were re-randomized to receive one of the two doses of elagolix (150 mg or 250 mg) QD for 12 weeks.
- Placebo / Elagolix 150 mg: Participants initially randomized to placebo were re-randomized at week 12 to receive elagolix 150 mg for 12 weeks.
- Placebo / Elagolix 250 mg: Participants initially randomized to placebo were re-randomized at week 12 to receive elagolix 250 mg for 12 weeks.
Period: Weeks 1 - 12
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg
Started | 52 | 51 | 52 | 0 | 0
Completed | 38 | 45 | 42 | 0 | 0
Not Completed | 14 | 6 | 10 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 4 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 2 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 0 | 0 | 0
Period: Weeks 13 - 24
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg
Started | 0 | 45 | 42 | 18 | 20
Completed | 0 | 38 | 37 | 14 | 18
Not Completed | 0 | 7 | 5 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 2 | 2
Not completed — Non-compliance | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Total
Number analyzed (Participants) | 52 | 51 | 52 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (1.0) | 30.9 (1.0) | 31.0 (1.0) | 31.0 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 52 | 155
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 2 | 2
  Black | 4 | 4 | 3 | 11
  White | 43 | 42 | 41 | 126
  Hispanic | 3 | 4 | 6 | 13
  Other | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Monthly Mean Numerical Rating Score (NRS) for Endometriosis Pain at Week 12
Description: The NRS is an 11-point scale used to measure endometriosis pain and was completed at approximately the same time each day using an electronic diary (e-Diary). Participants were instructed to select a single number between 0 (No pain) and 10 (Worst pain ever) that best described their endometriosis pain at its worst over the past day.
  The monthly mean NRS is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and week 12
Population: All randomized participants who received at least one dose of randomized, double-blind study drug and reported at least 10 e-Diary NRS values during the initial 12 week treatment period. The analysis includes participants with non-missing data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 38 | 44 | 45
units on a scale | -0.88 (0.18) | -1.19 (0.18) | -1.25 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Change from baseline in in monthly mean values of the NRS for overall endometriosis-associated pelvic pain was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.2311, Repeated Measures Analysis of Covariance; LS Mean Difference = -0.31, 95% CI 2-sided [-0.81 to 0.20], Standard Error of Mean 0.25 — Difference = Elagolix - Placebo
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1521, Repeated Measures Analysis of Covariance; LS Mean Difference = -0.36, 95% CI 2-sided [-0.86 to 0.14], Standard Error of Mean 0.25 — Difference = Elagolix - Placebo

2. Secondary Outcome: Change From Baseline in the Monthly Mean Numerical Rating Score (NRS) for Endometriosis Pain
Description: as for outcome 1
Time Frame: Baseline and weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4 | -0.60 (0.17) | -0.90 (0.17) | -0.83 (0.17)
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | -0.71 (0.18) | -1.23 (0.17) | -0.94 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 4. Change from baseline in in monthly mean values of the NRS for overall endometriosis-associated pelvic pain was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.2041, Repeated Measures ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.77 to 0.17], Standard Error of Mean 0.24 — Difference = Elagolix - Placebo
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3375, Repeated Measures ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.69 to 0.24], Standard Error of Mean 0.24 — Difference = Elagolix - Placebo
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 8. Change from baseline in in monthly mean values of the NRS for overall endometriosis-associated pelvic pain was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0354, Repeated Measures ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-1.01 to -0.04], Standard Error of Mean 0.25 — Difference = Elagolix - Placebo
Statistical Analysis 4: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.3618, Repeated Measures ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.71 to 0.26], Standard Error of Mean 0.25 — Difference = Elagolix - Placebo

3. Secondary Outcome: Change From Baseline in the Monthly Peak Numerical Rating Score (NRS) for Endometriosis Pain
Description: The NRS is an 11-point scale used to measure endometriosis pain and was completed at approximately the same time each day using an electronic diary (e-Diary). Participants were instructed to select a single number between 0 (No pain) and 10 (Worst pain ever) that best described their endometriosis pain at its worst over the past day.
  The monthly peak NRS is the maximum of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4 | -1.27 (0.32) | -1.39 (0.32) | -1.58 (0.32)
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | -1.25 (0.34) | -1.94 (0.33) | -2.41 (0.33)
  Week 12: number analyzed (Participants) | 38 | 44 | 45
  Week 12 | -1.30 (0.36) | -2.45 (0.34) | -2.74 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 4. Change from baseline in in monthly peak values of the NRS for overall endometriosis-associated pelvic pain was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.7990, Repeated Measures ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-1.01 to 0.78], Standard Error of Mean 0.46 — Difference = Elagolix - Placebo
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5042, Repeated Measures ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-1.21 to 0.59], Standard Error of Mean 0.46 — Difference = Elagolix - Placebo
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 8. Change from baseline in in monthly peak values of the NRS for overall endometriosis-associated pelvic pain was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.1459, Repeated Measures ANCOVA; LS Mean Difference = -0.69, 95% CI 2-sided [-1.63 to 0.24], Standard Error of Mean 0.48 — Difference = Elagolix - Placebo
Statistical Analysis 4: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0163, Repeated Measures ANCOVA; LS Mean Difference = -1.16, 95% CI 2-sided [-2.10 to -0.21], Standard Error of Mean 0.48 — Difference = Elagolix - Placebo
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 12. Change from baseline in in monthly peak values of the NRS for overall endometriosis-associated pelvic pain was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0207, Repeated Measures ANCOVA; LS Mean Difference = -1.15, 95% CI 2-sided [-2.13 to -0.18], Standard Error of Mean 0.50 — Difference = Elagolix - Placebo
Statistical Analysis 6: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0038, Repeated Measures ANCOVA; LS Mean Difference = -1.44, 95% CI 2-sided [-2.42 to -0.47], Standard Error of Mean 0.50 — Difference = Elagolix - Placebo

4. Secondary Outcome: Change From Baseline in the Monthly Mean Non-menstrual Pelvic Pain Score
Description: Participants assessed their pelvic pain not related to menses and its impact on their daily activities at approximately the same time every day in an e-Diary according to the following response options:
  * 0 = No pelvic pain
  * 1 = Mild pelvic pain; subject could not do some of the things she usually does
  * 2 = Moderate pelvic pain; subject could not do many of the things she usually does
  * 3 = Severe pelvic pain; subject could not do most or all of the things she usually does.
  The monthly mean non-menstrual pelvic pain score is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4 | -0.14 (0.05) | -0.18 (0.05) | -0.16 (0.05)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | -0.12 (0.05) | -0.30 (0.05) | -0.17 (0.05)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | -0.22 (0.06) | -0.27 (0.05) | -0.25 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 4. Change from baseline in non-menstrual pelvic pain score was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.5744, Repeated Measures ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.18 to 0.10], Standard Error of Mean 0.07 — Difference = Elagolix - Placebo
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7280, Repeated measures ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.17 to 0.12], Standard Error of Mean 0.07 — Difference = Elagolix - Placebo
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 8. Change from baseline in non-menstrual pelvic pain score was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0195, Repeated Measures ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.32 to -0.03], Standard Error of Mean 0.07 — Difference = Elagolix - Placebo
Statistical Analysis 4: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.5589, Repeated Measures ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.19 to 0.10], Standard Error of Mean 0.08 — Difference = Elagolix - Placebo
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 12. Change from baseline in non-menstrual pelvic pain score was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.5558, Repeated Measures ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.20 to 0.11], Standard Error of Mean 0.08 — Difference = Elagolix - Placebo
Statistical Analysis 6: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.7121, Repeated Measures ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.18 to 0.12], Standard Error of Mean 0.08 — Difference = Elagolix - Placebo

5. Secondary Outcome: Change From Baseline in the Monthly Mean Dysmenorrhea Score
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities at approximately the same time each day in an e-Diary according to the following response options:
  * Subject is not having her period
  * 0 = No pain related to period
  * 1 = Mild pain related to period; subject could not do some of the things she usually does
  * 2 = Moderate pain related to period; subject could not do many of the things she usually does
  * 3 = Severe pain related to period; subject could not do most of or all of the things she usually does.
  The monthly mean dysmenorrhea score is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4 | -0.20 (0.09) | -0.49 (0.09) | -0.40 (0.09)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | -0.29 (0.10) | -0.71 (0.09) | -0.79 (0.09)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | -0.24 (0.10) | -0.68 (0.10) | -0.76 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 4. Change from baseline in dysmenorrhea score was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0286, Repeated Measures ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.54 to -0.03], Standard Error of Mean 0.13 — Difference = Elagolix - Placebo
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1210, Repeated Measures ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.45 to 0.05], Standard Error of Mean 0.13 — Difference = Elagolix - Placebo
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 8. Change from baseline in dysmenorrhea score was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0024, Repeated Measures ANCOVA; LS Mean Difference = -0.42, 95% CI 2-sided [-0.68 to -0.15], Standard Error of Mean 0.14 — Difference = Elagolix - Placebo
Statistical Analysis 4: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0003, Repeated Measures ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.76 to -0.22], Standard Error of Mean 0.14 — Difference = Elagolix - Placebo
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 12. Change from baseline in dysmenorrhea score was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0021, Repeated Measures ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.72 to -0.16], Standard Error of Mean 0.14 — Difference = Elagolix - Placebo
Statistical Analysis 6: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0003, Repeated Measures ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.80 to -0.24], Standard Error of Mean 0.14 — Difference = Elagolix - Placebo

6. Secondary Outcome: Change From Baseline in the Monthly Mean Total of Dysmenorrhea and Non-menstrual Pelvic Pain Scores
Description: Participants assessed dysmenorrhea and pelvic pain not related to menses and their impact on daily activities at approximately the same time every day on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe) in an e-Diary.
  The sum of the dysmenorrhea and non-menstrual pelvic pain scores on each day were calculated to create a daily total score. On days the participant was not having her period, the dysmenorrhea score was not defined; hence, the total score was equal to the non-menstrual pelvic pain score (range 0 to 3). On days where the participant recorded menstruation the total score ranged from 0 to 6, where higher scores indicate more severe pain. The monthly mean sum of dysmenorrhea and non-menstrual pelvic pain scores is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4 | -0.18 (0.06) | -0.34 (0.06) | -0.29 (0.06)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | -0.18 (0.06) | -0.48 (0.06) | -0.33 (0.06)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | -0.27 (0.07) | -0.44 (0.06) | -0.41 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 4. Change from baseline in total of non-menstrual pelvic pain and dysmenorrhea scores was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0603, Repeated Measures ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.34 to 0.01], Standard Error of Mean 0.09 — Difference = Elagolix - Placebo
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.1855, Repeated Measures ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.29 to 0.06], Standard Error of Mean 0.09 — Difference = Elagolix - Placebo
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 8. Change from baseline in total of non-menstrual pelvic pain and dysmenorrhea scores was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0012, Repeated Measures ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.48 to -0.12], Standard Error of Mean 0.09 — Difference = Elagolix - Placebo
Statistical Analysis 4: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.1002, Repeated Measures ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.33 to 0.03], Standard Error of Mean 0.09 — Difference = Elagolix - Placebo
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg; Analysis at week 12. Change from baseline in total of non-menstrual pelvic pain and dysmenorrhea scores was analyzed by a repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for subject, and the baseline-by-time interaction, and the baseline value as a covariate; Test type: Superiority; p = 0.0568, Repeated Measures ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.36 to 0.01], Standard Error of Mean 0.09 — Difference = Elagolix - Placebo
Statistical Analysis 6: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.1190, Repeated Measures ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.33 to 0.04], Standard Error of Mean 0.09 — Difference = Elagolix - Placebo

7. Secondary Outcome: Percentage of Days With No Pain Based on NRS
Description: The NRS is an 11-point scale used to measure endometriosis pain and was completed at approximately the same time each day using an electronic diary (e-Diary). Participants were instructed to select a single number between 0 (No pain) and 10 (Worst pain ever) that best described their endometriosis pain at its worst over the past day.
  The percentage of days a participant reported a value of zero (or "no pain") for the NRS was calculated for the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Baseline | 27.600 (3.588) | 25.380 (3.564) | 25.515 (3.493)
  Week 4 | 35.252 (4.118) | 36.401 (4.606) | 32.355 (4.604)
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | 40.861 (4.671) | 43.780 (5.114) | 36.737 (5.467)
  Week 12: number analyzed (Participants) | 38 | 44 | 45
  Week 12 | 47.431 (4.955) | 44.841 (5.857) | 41.760 (5.796)

8. Secondary Outcome: Percentage of Days With No Pain Based Based on Non-menstrual Pelvic Pain Daily Assessment
Description: Participants assessed their pelvic pain not related to menses and its impact on their daily activities at approximately the same time every day in an e-Diary according to the following response options:
  * 0 = No pelvic pain
  * 1 = Mild pelvic pain; subject could not do some of the things she usually does
  * 2 = Moderate pelvic pain; subject could not do many of the things she usually does
  * 3 = Severe pelvic pain; subject could not do most or all of the things she usually does.
  The percentage of days a participant reported a value of zero ("no pain") for non-menstrual pelvic pain was calculated for the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Baseline | 34.939 (3.831) | 36.821 (4.041) | 38.530 (4.065)
  Week 4 | 42.986 (4.229) | 45.469 (4.968) | 44.443 (4.905)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | 46.228 (4.777) | 54.967 (5.291) | 47.524 (5.367)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | 54.270 (4.768) | 53.836 (6.077) | 50.061 (5.496)

9. Secondary Outcome: Percentage of Days With No Pain Based Based on Dysmenorrhea Daily Assessment
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities at approximately the same time each day in an e-Diary according to the following response options:
  * Subject is not having her period
  * 0 = No pain related to period
  * 1 = Mild pain related to period; subject could not do some of the things she usually does
  * 2 = Moderate pain related to period; subject could not do many of the things she usually does
  * = Severe pain related to period; subject could not do most of or all of the things she usually does.
  The percentage of days a participant reported a value of zero ("no pain") for dysmenorrhea was calculated for the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Baseline | 26.350 (3.710) | 14.340 (2.154) | 21.086 (3.210)
  Week 4 | 30.513 (4.435) | 43.411 (5.775) | 39.475 (5.509)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | 35.057 (5.135) | 56.952 (6.016) | 67.411 (6.190)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | 34.439 (5.000) | 61.658 (6.717) | 66.186 (6.336)

10. Secondary Outcome: Percentage of Days With No Pain Based Based on Total Score of Non-menstrual Pelvic Pain and Dysmenorrhea Daily Assessment
Description: Participants assessed dysmenorrhea and pelvic pain not related to menses and their impact on daily activities at approximately the same time every day in an e-Diary on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe). The sum of the dysmenorrhea and non-menstrual pelvic pain scores on each day were calculated to create a daily total score. On days the participant was not having her period, the dysmenorrhea score was not defined; hence, the total score was equal to the non-menstrual pelvic pain score (range 0 to 3). On days where the participant recorded menstruation the total score ranged from 0 to 6, where higher scores indicate more severe pain.
  The percentage of days a participant reported a value of zero ("no pain") for the non-menstrual pelvic pain and dysmenorrhea total score was calculated for the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Baseline | 33.009 (3.690) | 32.940 (3.649) | 35.967 (3.815)
  Week 4 | 39.586 (4.058) | 44.020 (4.825) | 43.230 (4.844)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | 43.961 (4.607) | 53.526 (5.200) | 47.108 (5.380)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | 50.340 (4.552) | 52.584 (5.999) | 49.409 (5.494)

11. Secondary Outcome: Change From Baseline in the Percentage of Days of Any Analgesic Use
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of any analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of an analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Week 4 | -4.8 (2.3) | -8.7 (2.3) | -6.8 (2.3)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | -5.8 (2.4) | -12.6 (2.4) | -10.4 (2.4)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | -6.1 (2.5) | -10.5 (2.4) | -13.9 (2.4)

12. Secondary Outcome: Change From Baseline in the Percentage of Days of Prescription Analgesic Use
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of prescription analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of a prescription analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Week 4 | -1.0 (1.2) | -4.0 (1.2) | -2.3 (1.2)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | -0.8 (1.4) | -3.2 (1.3) | -3.2 (1.4)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | -2.1 (1.6) | -2.6 (1.6) | -3.3 (1.6)

13. Secondary Outcome: Change From Baseline in the Percentage of Days of Narcotic Analgesic Use
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of narcotic analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of a narcotic analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of days
  Week 4 | -0.8 (1.1) | -2.5 (1.2) | -2.1 (1.2)
  Week 8: number analyzed (Participants) | 45 | 48 | 47
  Week 8 | -0.8 (1.2) | -1.8 (1.2) | -3.0 (1.2)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | -1.7 (1.3) | -1.3 (1.3) | -3.6 (1.3)

14. Secondary Outcome: Percentage of Participants With 30% Decrease From Baseline in Monthly Mean NRS
Description: as for outcome 1
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants
  Week 4 | 38.5 [25.2 to 51.7] | 43.1 [29.5 to 56.7] | 47.1 [33.4 to 60.8]
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | 54.5 [39.8 to 69.3] | 60.4 [46.6 to 74.3] | 51.1 [36.8 to 65.4]
  Week 12: number analyzed (Participants) | 38 | 44 | 45
  Week 12 | 60.5 [45.0 to 76.1] | 63.6 [49.4 to 77.9] | 60.0 [45.7 to 74.3]

15. Secondary Outcome: Percentage of Participants With 30% Decrease From Baseline in Monthly Peak NRS
Description: as for outcome 3
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants
  Week 4 | 30.8 [18.2 to 43.3] | 35.3 [22.2 to 48.4] | 31.4 [18.6 to 44.1]
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | 38.6 [24.2 to 53.0] | 43.8 [29.7 to 57.8] | 48.9 [34.6 to 63.2]
  Week 12: number analyzed (Participants) | 38 | 44 | 45
  Week 12 | 36.8 [21.5 to 52.2] | 47.7 [33.3 to 62.5] | 57.8 [43.3 to 72.2]

16. Secondary Outcome: Percentage of Participants With 50% Decrease From Baseline in Monthly Mean NRS
Description: as for outcome 1
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants
  Week 4 | 21.2 [10.1 to 32.3] | 37.3 [24.0 to 50.5] | 25.5 [13.5 to 37.5]
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | 36.4 [22.1 to 50.6] | 45.8 [31.7 to 59.9] | 38.3 [24.4 to 52.2]
  Week 12: number analyzed (Participants) | 38 | 44 | 45
  Week 12 | 36.8 [21.5 to 52.2] | 45.5 [30.7 to 60.2] | 44.4 [29.9 to 59.0]

17. Secondary Outcome: Percentage of Participants With 50% Decrease From Baseline in Monthly Peak NRS
Description: as for outcome 3
Time Frame: Baseline and weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants
  Week 4 | 11.5 [2.9 to 20.2] | 17.6 [7.2 to 28.1] | 19.6 [8.7 to 30.5]
  Week 8: number analyzed (Participants) | 44 | 48 | 47
  Week 8 | 11.4 [2.0 to 20.7] | 25.0 [12.8 to 37.2] | 36.2 [22.4 to 49.9]
  Week 12: number analyzed (Participants) | 38 | 44 | 45
  Week 12 | 23.7 [10.2 to 37.2] | 34.1 [20.1 to 48.1] | 42.2 [27.8 to 56.7]

18. Secondary Outcome: Change From Baseline in Dyspareunia Component of the Composite Pelvic Signs and Symptoms Score (CPSSS)
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. To assess dyspareunia (painful intercourse) participants were asked to select the best description of pain during sexual intercourse over the past 28 days using the following response categories:
  * 0 = Absent; No discomfort during sexual intercourse.
  * 1 = Mild; I can tolerate the discomfort during sexual intercourse.
  * 2 = Moderate; Intercourse is sometime interrupted due to pain.
  * 3 = Severe; I prefer to avoid intercourse because of pain.
  * Not applicable. I am not sexually active for reasons other than my endometriosis symptoms.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4: number analyzed (Participants) | 37 | 37 | 31
  Week 4 | -0.19 (0.12) | -0.21 (0.12) | -0.56 (0.13)
  Week 8: number analyzed (Participants) | 34 | 37 | 25
  Week 8 | -0.15 (0.12) | -0.68 (0.12) | -0.66 (0.14)
  Week 12: number analyzed (Participants) | 32 | 35 | 28
  Week 12 | -0.29 (0.13) | -0.67 (0.12) | -0.49 (0.14)

19. Secondary Outcome: Patient Global Impression of Change at Weeks 4, 8 and 12
Description: The Patient Global Impression of Change (PGIC) is a questionnaire-based assessment of the change in endometriosis pain since the initiation of study drug. The participant was asked to select from one of seven response categories:
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. Not Changed
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Week 4: number analyzed (Participants) | 48 | 50 | 50
  Week 4 | 3.4 (0.2) | 3.0 (0.2) | 2.8 (0.2)
  Week 8: number analyzed (Participants) | 46 | 48 | 45
  Week 8 | 3.0 (0.2) | 2.3 (0.1) | 2.4 (0.2)
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | 3.2 (0.2) | 2.2 (0.2) | 2.2 (0.2)

20. Secondary Outcome: Percentage of Participants With a PGIC Response of Minimally Improved, Much Improved, or Very Much Improved
Description: as for outcome 19
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants
  Week 4: number analyzed (Participants) | 48 | 50 | 50
  Week 4 | 54.2 [40.1 to 68.3] | 62.0 [48.5 to 75.5] | 80.0 [68.9 to 91.1]
  Week 8: number analyzed (Participants) | 46 | 48 | 45
  Week 8 | 67.4 [53.8 to 80.9] | 91.7 [83.8 to 99.5] | 84.4 [73.9 to 95.0]
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | 60.0 [44.8 to 75.2] | 88.9 [79.7 to 98.1] | 82.2 [71.1 to 93.4]

21. Secondary Outcome: Percentage of Participants With a PGIC Response of Much Improved or Very Much Improved
Description: as for outcome 19
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants
  Week 4: number analyzed (Participants) | 48 | 50 | 50
  Week 4 | 12.5 [3.1 to 21.9] | 34.0 [20.9 to 47.1] | 38.0 [24.5 to 51.5]
  Week 8: number analyzed (Participants) | 46 | 48 | 45
  Week 8 | 37.0 [23.0 to 50.9] | 58.3 [44.4 to 72.3] | 60.0 [45.7 to 74.3]
  Week 12: number analyzed (Participants) | 40 | 45 | 45
  Week 12 | 32.5 [18.0 to 47.0] | 66.7 [52.9 to 80.4] | 62.2 [48.1 to 76.4]

22. Secondary Outcome: Change From Baseline in Endometriosis Health Profile-5 (EHP-5) at Week 12
Description: The EHP-5 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-5 consists of two parts:
  * A core questionnaire consisting of five questions that measure the areas of pain, control and powerlessness, emotional well-being, social support, and self-image with five response categories for each item (Never, Rarely, Sometimes, Often, Always)
  * A supplemental questionnaire consisting of six additional questions which assess the areas of work, relationship with children, sexual intercourse, feelings about the medical profession, treatment, and infertility with the same five response categories plus an additional response category of Not Relevant which was not scored.
  The scores associated with each possible outcome category are as follows: never (0), rarely (25), sometimes (50), often (75), and always (100). A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 52 | 51 | 51
units on a scale
  Pain: number analyzed (Participants) | 38 | 45 | 42
  Pain | -11.8 (3.6) | -25.0 (3.3) | -17.3 (4.0)
  Control and Powerlessness: number analyzed (Participants) | 38 | 45 | 42
  Control and Powerlessness | -10.5 (4.7) | -25.6 (3.4) | -22.6 (4.8)
  Emotional Wellbeing: number analyzed (Participants) | 38 | 45 | 42
  Emotional Wellbeing | -6.6 (4.0) | -17.2 (3.5) | -9.5 (4.8)
  Social Support: number analyzed (Participants) | 38 | 45 | 42
  Social Support | -18.4 (4.2) | -25.0 (4.1) | -15.5 (4.8)
  Self-image: number analyzed (Participants) | 38 | 45 | 42
  Self-image | -9.9 (3.1) | -18.9 (3.7) | -10.7 (4.0)
  Work: number analyzed (Participants) | 36 | 40 | 35
  Work | -6.9 (4.2) | -28.8 (3.9) | -22.1 (3.2)
  Relationship with Children: number analyzed (Participants) | 25 | 27 | 16
  Relationship with Children | -7.0 (5.3) | -25.0 (4.4) | -20.3 (5.2)
  Sexual Intercourse: number analyzed (Participants) | 33 | 39 | 28
  Sexual Intercourse | -9.8 (4.6) | -23.1 (3.9) | -19.6 (5.5)
  Medical Profession: number analyzed (Participants) | 32 | 40 | 34
  Medical Profession | 0.0 (3.7) | -17.5 (3.9) | -14.0 (4.2)
  Frustration with Treatment: number analyzed (Participants) | 38 | 42 | 41
  Frustration with Treatment | -8.6 (4.7) | -26.2 (4.2) | -23.2 (5.4)
  Concerns with Infertility: number analyzed (Participants) | 28 | 34 | 33
  Concerns with Infertility | -9.8 (4.1) | -5.1 (4.1) | -9.1 (4.0)

23. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femur at Week 12
Description: Bone mineral density (BMD) of the femur (total hip) was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and week 12
Population: All randomized participants who received at least one dose of randomized, double-blind study drug and with available BMD data at baseline and week 12.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 37 | 42 | 43
percent change | -0.283 (1.851) | -0.294 (1.762) | -0.382 (1.338)

24. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femur at Week 24
Description: Bone mineral density (BMD) of the femur (total hip) was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of randomized, double-blind study drug and with available BMD data at baseline and week 24.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg
Number analyzed (Participants) | 37 | 37 | 13 | 17
percent change | -0.743 (1.877) | -1.024 (1.759) | -0.924 (1.198) | -0.076 (2.362)

25. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Spine at Week 12
Description: Bone mineral density (BMD) of the spine was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and week 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
Number analyzed (Participants) | 36 | 43 | 42
percent change | 0.375 (2.091) | -0.045 (2.088) | -0.937 (2.747)

26. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Spine at Week 24
Description: Bone mineral density (BMD) of the spine was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Week 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg
Number analyzed (Participants) | 38 | 37 | 14 | 15
percent change | -1.032 (1.983) | -1.631 (2.874) | -0.692 (1.724) | 0.681 (2.720)

ADVERSE EVENTS:
Time Frame: From the first dose of any study drug through week 24. The Placebo treatment group includes data for the initial 12-week treatment phase. The Elagolix treatment groups include data for the total 24-week treatment period for participants initially randomized to elagolix, and 12-week treatment period for participants initially randomized to placebo and re-randomized at week 12.
Groups:
- Placebo: Participants received elagolix 150 mg tablets once a day for 12 weeks.
- Elagolix 150 mg: Participants initially randomized to elagolix 150 mg received elagolix 150 mg tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 150 mg for an additional 12 weeks.
  Participants initially randomized to placebo were re-randomized at week 12 to receive elagolix 150 mg for 12 weeks.
- Elagolix 250 mg: Participants initially randomized to elagolix 250 mg received elagolix 250 mg tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 250 mg for an additional 12 weeks.
  Participants initially randomized to placebo were re-randomized at week 12 to receive elagolix 250 mg for 12 weeks.
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/69 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/69 | 1/72
Other Adverse Events (participants affected / at risk) | 18/52 | 31/69 | 33/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | Elagolix 150 mg (N=69) | Elagolix 250 mg (N=72)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | Elagolix 150 mg (N=69) | Elagolix 250 mg (N=72)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 6 (7) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 2 (4) | 3 (4)
SINUSITIS (Infections and infestations) | 2 (2) | 6 (6) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 6 (6) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 5 (5) | 4 (4)
VAGINAL MYCOSIS (Infections and infestations) | 3 (3) | 1 (1) | 6 (8)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 4 (4) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 6 (9) | 4 (12)
MIGRAINE (Nervous system disorders) | 0 (0) | 3 (3) | 4 (4)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.